CLINICAL TRIAL: NCT02687919
Title: Randomized Control Trial Evaluation of a Modified Paleolithic Dietary Intervention in the Treatment of Relapsing-Remitting Multiple Sclerosis: A Pilot Study
Brief Title: Evaluation of a Modified Paleolithic Dietary Intervention in the Treatment of Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amanda Irish (Other)
Responsible Party: Sponsor-Investigator, Amanda Irish, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201208703
Record Dates: First submitted 2016-01-22; First posted 2016-02-22 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: diet (gluten-free); diet therapy; quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Paleo Diet Intervention (MPDI) (Experimental): Consumed a modified Paleo diet, described as nine cups of vegetables and some fruits, meat protein including organ meat, and complete abstinence from products containing gluten (wheat, barley, rye, etc.), dairy, potatoes, and legumes (beans, lentils, peanuts, soy, etc.)
  Interventions: Other: Modified Paleo diet
- Usual Care (No Intervention): Typical physician recommendations for MS.

INTERVENTIONS:
Other: Modified Paleo diet — Nine cups of vegetables and some fruits, meat protein including organ meat, and complete abstinence from products containing gluten (wheat, barley, rye, etc.), dairy, potatoes, and legumes (beans, lentils, peanuts, soy, etc.)
  Other Names: Modified Paleolithic Diet
  Arms: Modified Paleo Diet Intervention (MPDI)

SUMMARY:
This is a research study. The investigators are inviting participants to participate in this research study between the ages of 18-45, who have stable Relapsing-Remitting Multiple Sclerosis (RRMS), are able to walk 25 ft with/without an assistive device, and have none of the following: liver disease, kidney disease, diabetes, active heart disease, heart block or arrhythmias, bleeding disorders, concurrent diuretic use, anti-coagulation or anti-platelet use, psychosis or other psychiatric disorder likely to impact ability to comply with study procedures, any change in prescription medication for a mental health problem such as depression or anxiety in the last three months.

The purpose of this research study is to determine whether or not a modified Paleolithic diet results in any change in health in persons with RRMS compared to usual care. The investigators define usual care as the typical or usual physician recommendations for the treatment of RRMS.

The Paleolithic diet (or Paleo diet), also referred to as the caveman diet, Stone Age diet, and hunter-gatherer diet, is a modern nutritional plan based on the presumed ancient diet of wild plants and animals of ancestral humans during the Paleolithic era (a period of about 2.5 million years duration that ended around 10,000 years ago with the development of agriculture). The diet consists mainly of fish, grass-fed pasture raised meats, vegetables, fruit, fungi, roots, and nuts, and excludes grains, legumes, dairy products, salt, refined sugar, and processed oils.

To the investigators' knowledge, most neurologists prescribe medications that may reduce or prevent future disability, but few prescribe dietary modifications unless needed for other concomitant disease.

DETAILED DESCRIPTION:
Initial visit/baseline measures for intervention and control groups (1-2 hrs): Subject Info and Demographics, Fatigue Severity Scale (FSS), Blood draw (vitamin B-1 (thiamine), vitamin B-9 (folate), vitamin B-12 (cobalamin), vitamin K, homocysteine, C-reactive protein), MS Functional Composite (MSFC) [Timed 25-Foot Walk (T25-FW), 9-Hole Peg Test (9-HPT), Paced Auditory Serial Addition Test (PASAT)], 6-minute walk, and Paced Visual Serial Addition Test (PVSAT).

Complete at home/office/other: Automated Self-Administered 24-hour recall application (ASA24).

Two-week run-in for intervention and control groups: Return survey instruments: [Multiple Sclerosis Quality of Life-54 (MSQOL-54), Veterans Specific Activity Questionnaire (VSAQ), Medication, Vitamin, and Supplement Log, and Food Diary]. Randomization; training for intervention and control groups (1-2 hrs). Training for the intervention group will involve orientation of subjects to the modified paleo diet and food logging; control group training will consist of study expectations (maintenance of normal diet) and food logging. Both will be conducted by a research team member, with subjects, on an individual basis.

Begin 3-month study: 1 short follow-up call per week, for first three weeks, then every other week thereafter asking intervention and control group subjects if they need assistance with study procedures and providing assistance when needed/possible and ensuring subjects are accurately maintaining daily food log/diary (5 mins; could be longer/shorter depending on subject needs). If a subject (intervention or control arm) is having difficulty filling out the Food Log/Food Diary, he/she will have the opportunity to meet with research team members at a location of the subject's choosing (to include web-conferencing) for supplemental instruction.

At 1 month and few days before returning for the final visit, complete at home/office/other: Automated Self-Administered 24-hour recall application (ASA24).

Final visit* for intervention and control groups (1-2 hrs): Multiple Sclerosis Quality of Life-54 (MSQOL-54), Fatigue Severity Scale (FSS), Veterans Specific Activity Questionnaire (VSAQ), Medication, Vitamin, and Supplement Log, Food Log, Blood draw (vitamin B-1 (thiamine), vitamin B-9 (folate), vitamin B-12 (cobalamin), vitamin K, homocysteine, C-reactive protein), MS Functional Composite (MSFC) [Timed 25-Foot Walk (T25-FW), 9-Hole Peg Test (9-HPT), Paced Auditory Serial Addition Test (PASAT)], 6-minute walk, and Paced Visual Serial Addition Test (PVSAT). *End of participation for intervention group or cross-over (from control to 3-month intervention) for interested control group subjects.

If regular in-person meetings are not possible (for two-week recall and/or supplemental instruction), a subject may choose to communicate with research staff via a web conferencing application (Google Hangout). The privacy policy may be found here: http://www.google.com/policies/privacy/ and will be provided to subjects upon request.

ELIGIBILITY:
Inclusion Criteria:

1. Verified diagnosis of relapsing-remitting multiple sclerosis (RRMS) with no change in medications in the prior three months.
2. Able to ambulate a minimum of 25 feet with/without use of an assistive device.

Exclusion Criteria:

1. Under the age of 18 or over the age of 45 at the beginning of the study.
2. Unstable MS, requiring a change in medication in the prior 3 months.
3. Unwillingness to contact, or allow research to contact, neurologist for verification of RRMS diagnosis.
4. Psychosis or other psychiatric disorder likely to impact ability to comply with study procedures.
5. Change in prescriptions medication in the prior three months for a mental health problem such as depression or anxiety.
6. Active malignancy undergoing treatment (not including non melanoma skin cancers).
7. Subjects with liver disease, kidney disease, diabetes, active heart disease, heart block or arrhythmias, bleeding disorders, concurrent diuretic use, anti-coagulation or anti-platelet use.
8. Abnormal bleeding disorder.
9. On any "diet" recommended to treat MS (ex: Best Bet, Swank, McDougall, MS Recovery diet, Wahls', other Paleolithic, gluten-free, vegetarian, and/or vegan
10. Inability to maintain food log for for seven consecutive days during the run-in phase of the study.
11. Not comfortable using a computer.
12. Other failure to demonstrate compliance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K Irish, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study are complex and housed in different formats, but are available by contacting the corresponding author.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Started | 16 | 15
Completed | 8 | 9
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (5.7) | 37.1 (3.7) | 36.2 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 1 | 1 | 2
Fatigue Severity Scale (FSS)-9 [Mean (Standard Deviation); unit: units on a scale] — Higher score (1-7) indicates more fatigue. The total score is the average of 9 questions.
  units on a scale | 4.2 (1.6) | 4.0 (1.2) | 4.1 (1.4)
Veterans Specific Activity Questionnaire (VSAQ) [Mean (Standard Deviation); unit: units on a scale] — Estimates exercise tolerance in metabolic equivalents (METs). A higher score (1-13) indicates better exercise tolerance.
  units on a scale | 6.1 (2.4) | 5.8 (2.5) | 6.0 (2.4)
Timed 25-Foot Walk (25-FW) [Mean (Standard Deviation); unit: seconds] — Quantitative mobility and leg function performance test based on a timed 25-foot walk. Less time to complete indicates less physical fatigue.
  seconds | 4.7 (0.7) | 4.7 (0.5) | 4.7 (0.6)
9-Hole Peg Test (9-HPT) (dominant) [Mean (Standard Deviation); unit: seconds] — On a start command, a stopwatch is started, the patient picks up nine pegs one at-a-time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at-a-time, replacing them into the shallow container. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged.
  seconds | 21.0 (3.9) | 19.6 (2.0) | 20.3 (3.1)
9-Hole Peg Test (9-HPT) (nondominant) [Mean (Standard Deviation); unit: seconds] — On a start command, a stopwatch is started, the patient picks up nine pegs one at-a-time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at-a-time, replacing them into the shallow container. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged.
  seconds | 24.4 (4.5) | 20.4 (3.6) | 22.4 (4.4)
Paced Auditory Serial Addition Test (PASAT) [Mean (Standard Deviation); unit: units on a scale] — Total number correct out of 60 possible answers. A higher score indicates reduced cognitive fatigue.
  units on a scale | 44.9 (4.5) | 53.2 (5.0) | 49 (6.3)
6 Minute Walk (6-MW) [Mean (Standard Deviation); unit: meters] — Assesses submaximal aerobic capacity/endurance through measuring distance walked in 6 minutes. Greater distance indicates less physical fatigue.
  meters | 570.1 (56.0) | 532.9 (56.1) | 551.5 (57.5)
Multiple Sclerosis Quality of Life-54 (MSQOL-54) (physical) [Mean (Standard Deviation); unit: units on a scale] — This 54-item instrument generates two composite summary scores, physical health and mental health. Higher scores (0-100) indicate improved health.
  units on a scale | 67.3 (15.2) | 68.1 (11.8) | 67.7 (13.1)
Multiple Sclerosis Quality of Life-54 (MSQOL-54) (mental) [Mean (Standard Deviation); unit: units on a scale] — This 54-item instrument generates two composite summary scores, physical health and mental health. Higher scores (0-100) indicate improved health.
  units on a scale | 74.5 (10.8) | 65.5 (11.5) | 70 (11.8)
B-1 (thiamine) [Mean (Standard Deviation); unit: nmol/L] | 150.8 (28.7) | 129.5 (36.0) | 140.1 (33.3)
B-9 (folate) [Mean (Standard Deviation); unit: ng/mL] — Population: One sample from usual care was lost.
  ng/mL
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 15.68 (2.01) | 17.51 (1.2) | 16.06 (4.53)
B-12 (cobalamin) [Mean (Standard Deviation); unit: pg/mL] | 663.1 (183.6) | 498.0 (153.0) | 580.5 (183.5)
K (pg/mL) [Mean (Standard Deviation); unit: pg/mL] | 1643.4 (863.3) | 1758.3 (910.6) | 1700.8 (859.2)
HCY [Mean (Standard Deviation); unit: μmol/L] | 9.4 (1.8) | 9.3 (3.7) | 9.3 (3.0)
Hs-CRP [Mean (Standard Deviation); unit: mg/L] | 4.4 (4.3) | 1.4 (1.2) | 2.9 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue Severity Scale (FSS)-9 Score
Description: Specific Aims: 1) Test the hypothesis that a modified Paleolithic diet reduces effects of fatigue in subjects with Relapsing-Remitting Multiple Sclerosis (RRMS), compared to controls, in: (a) daily life as measured by the Fatigue Severity Scale (FSS) score.
  A 9-item sel-report questionnaire related to how fatigue interferes with certain activities and rates its severity, items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score is 9 and maximum score is 63. Higher the score indicates greater fatigue severity.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
units on a scale
  Baseline | 4.20 (0.60) | 3.99 (0.43)
  End of study | 2.82 (0.51) | 4.25 (0.43)

2. Primary Outcome: Change in Paced Auditory Serial Addition Test (PASAT) Score
Description: Specific Aims: 1) Test the hypothesis that a modified Paleolithic diet reduces effects of fatigue in subjects with Relapsing-Remitting Multiple Sclerosis (RRMS), compared to controls, in: (b) cognitive fatigue as measured by the Paced Auditory Serial Addition Test (PASAT) score.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio to ensure standardization in the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The score for the PASAT (0-60) is the total number correct out of 60 possible answers.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
units on a scale
  Baseline | 44.88 (1.71) | 53.22 (1.78)
  End of Study | 49.75 (2.66) | 54.89 (1.30)

3. Primary Outcome: Change in 6-minute Walk (6-MW) Distance
Description: Specific Aims: 1) Test the hypothesis that a modified Paleolithic diet reduces effects of fatigue in subjects with Relapsing-Remitting Multiple Sclerosis (RRMS), compared to controls, in: (c) physical fatigue as measured by the 6-minute (m) walk (6-MW).
  Timed 6-minute walk (6-MW): a submaximal measure of gait velocity and endurance over a distance (m) walked in 6 minutes.
Time Frame: End of Study, 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: meters
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
meters
  Baseline | 570.11 (21.15) | 532.95 (19.85)
  End of Study | 631.14 (12.30) | 562.47 (29.53)

4. Primary Outcome: Change in (25-FW) 25-ft Walk Time
Description: Specific Aims: 1) Test the hypothesis that a modified Paleolithic diet reduces effects of fatigue in subjects with Relapsing-Remitting Multiple Sclerosis (RRMS), compared to controls, in: (d) physical fatigue as measured by the 25-ft walk (25-FW; (s).
  Timed 25-Foot Walk (T25-FW): a quantitative test of maximal walking velocity, mobility, dynamic balance and leg function. The subject is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly and as safely, as possible. The time is recorded from the first step across the line and ends when the patient crosses the same foot over the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
Seconds
  Baseline | 4.67 (0.27) | 4.65 (0.18)
  End of study | 4.13 (0.20) | 4.51 (0.20)

5. Secondary Outcome: Quality of Life (MSQOL-54)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by: Multiple Sclerosis Quality of Life-54 (MSQOL-54) Mental and Physical Health scores.
  Multiple Sclerosis Quality of Life-54 (MSQOL-54): a multidimensional health-related quality of life survey that combines both generic and MS-specific items into a single instrument. Higher scores (0-100) indicate improved health.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
units on a scale
  Physical Baseline | 67.26 (5.76) | 68.08 (4.17)
  Mental Baseline | 74.47 (4.07) | 65.46 (4.07)
  Physical End of Study | 81.77 (3.51) | 65.62 (2.77)
  Mental End of Study | 86.53 (3.51) | 64.51 (4.65)

6. Secondary Outcome: Quality of Life (Vitamin B-1 Blood Serum Measures)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by vitamin B-1 (thiamine) blood serum measures.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: units listed
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
units listed
  B-1 (nmol/L) Baseline | 150.75 (10.85) | 129.50 (12.74)
  B-1 (nmol/L) End of Study | 146.13 (21.78) | 127.11 (15.43)

7. Secondary Outcome: Quality of Life (Vitamin B-9 Blood Serum Measures)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by vitamin B-9 (folate) blood serum measures.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Population: One baseline sample from usual care was lost.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
ng/mL
  B-9 (ng/mL) Baseline: number analyzed (Participants) | 8 | 8
  B-9 (ng/mL) Baseline | 15.68 (2.01) | 17.51 (1.12)
  B-9 (ng/mL) End of Study | 15.61 (1.99) | 17.43 (1.2)

8. Secondary Outcome: Quality of Life (Vitamins B-12 and K Blood Serum Measures)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by blood serum measures: vitamin B-12 (cobalamin) and vitamin K.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
pg/mL
  B-12 (pg/mL) Baseline | 663.14 (69.40) | 497.96 (54.09)
  K (pg/mL) Baseline | 1643.38 (326.28) | 1758.25 (321.94)
  B-12 (pg/mL) End of Study | 638.93 (75.27) | 500.21 (47.67)
  K (pg/mL) End of Study | 5949.63 (2100.8) | 1694.78 (518.94)

9. Secondary Outcome: Quality of Life (Homocysteine Blood Serum Measures)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by homocysteine (HCY) blood serum measures.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: μmol/L
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
μmol/L
  HCY (μmol/L) Baseline | 9.37 (0.70) | 9.27 (1.33)
  HCY (μmol/L) End of Study | 9.66 (0.94) | 10.01 (1.57)

10. Secondary Outcome: Quality of Life (C-reactive Protein Blood Serum Measures)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by C-reactive protein (hs-CRP) blood serum measures.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 9 | 9
mg/L
  Hs-CRP (mg/L) Baseline | 4.35 (1.64) | 1.40 (0.44)
  Hs-CRP (mg/L) End of Study | 3.26 (1.75) | 1.93 (0.52)

11. Secondary Outcome: Quality of Life (9-HPT)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by the 9-Hole Peg Test (9-HPT).
  9-Hole Peg Test: a brief, standardized, quantitative test of upper extremity function. The patient is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes (Rolyan 9-Hole Peg Test Kit - Model A8515). On a start command a stopwatch is started, the patient picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The score for the 9-HPT is an average of the two trials for each hand.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
seconds
  Dominant Baseline | 20.98 (1.49) | 19.61 (0.72)
  Non-dominant Baseline | 24.36 (1.70) | 20.41 (1.26)
  Dominant End of Study | 17.81 (0.88) | 19.02 (0.58)
  Non-dominant End of Study | 19.93 (1.23) | 18.89 (0.86)

12. Secondary Outcome: Quality of Life (VSAQ)
Description: Test the hypothesis that a modified Paleolithic diet improves general well-being/health and quality of life of RRMS patients, compared to controls, as measured by the Veterans Specific Activity Questionnaire (VSAQ).
  Veterans Specific Activity Questionnaire (VSAQ): a self-reported survey instrument that serves as a strong predictor of both measured and predicted exercise capacity. Subjects identify a series of activities that they can complete on a typical day (scaled 1-11 for estimated metabolic equivalents (METs)), higher METs indicate increased exercise capacity.
Time Frame: End of Study, measured at 3.5 months; Change from Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
Number analyzed (Participants) | 8 | 9
units on a scale
  Baseline | 6.13 (0.91) | 5.78 (0.88)
  End of Study | 7.75 (0.98) | 5.78 (0.84)

ADVERSE EVENTS:
Time Frame: Length of participant involvement (3.5 mos or 6.5 mos for cross-over subjects).
Description: No adverse events were reported by subjects.
Arm/Group | Modified Paleo Diet Intervention (MPDI) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No